CLINICAL TRIAL: NCT00111124
Title: Enbrel® in Psoriatic Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 20030106
Record Dates: First submitted 2005-05-17; First posted 2005-05-18 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Psoriasis
Keywords: psoriasis; arthritis; Enbrel®; etanercept
MeSH Terms: conditions — Psoriasis; Arthritis | interventions — Etanercept

INTERVENTIONS:
Drug: Enbrel®

SUMMARY:
This study is testing the effect of etanercept in treating both the skin and joint symptoms of psoriatic arthritis patients. Enbrel®, also known as etanercept, has already been approved by the Federal Food Drug Administration for the treatment of psoriatic arthritis. It is taken as an injection under the skin. Participants in the trial will be offered etanercept free of charge to be self-injected once weekly for 24 weeks. During that period they will have 5 appointments at the study center and will also be asked to complete assessments of their health.

ELIGIBILITY:
Individuals may be eligible to enroll in this study if they suffer from psoriasis (covering at least 10% of the body), and: - have had two or more swollen, tender or painful joints for at least 3 months or: - have lower back pain which your physician has diagnosed as sacroiliitis or spondylitis in one or more joints or: - have been diagnosed with active psoriatic arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
The proportion of subjects achieving a status on the Physician Global Assessment of Psoriasis of ""mild"" or better at week 24.

SECONDARY OUTCOMES:
Quality of life and disability as measured by the DLQI and HAQ
Financial impact of therapy on disease as measured by Patient Pharmacoeconomic Questionnaire
Serious Adverse Events
Patient Global Assessment of Psoriasis
Patient Global Assessment of Joint Disease
Patient Global Assessment of Joint Pain
Patient Assessment of Morning Stiffness Duration

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Frankel EH, Strober BE, Crowley JJ, Fivenson DP, Woolley JM, Yu EB, Xia HA, Chiou CF, Stevens SR. Etanercept improves psoriatic arthritis patient-reported outcomes: results from EDUCATE. Cutis. 2007 Apr;79(4):322-6. PMID 17500381
- [Result] Gottlieb AB, Kircik L, Eisen D, Jackson JM, Boh EE, Strober BE, Frankel E, Xia HA, Stevens SR. Use of etanercept for psoriatic arthritis in the dermatology clinic: the Experience Diagnosing, Understanding Care, and Treatment with Etanercept (EDUCATE) study. J Dermatolog Treat. 2006;17(6):343-52. doi: 10.1080/09546630600967166. PMID 17853307
- [Result] Gottlieb AB, Mease PJ, Mark Jackson J, Eisen D, Amy Xia H, Asare C, Stevens SR. Clinical characteristics of psoriatic arthritis and psoriasis in dermatologists' offices. J Dermatolog Treat. 2006;17(5):279-87. doi: 10.1080/09546630600823369. PMID 17092858
- [Result] Kimball AB, Jackson JM, Sobell JM, Boh EE, Grekin S, Pharmd EB, Woolley JM, Xia HA, Chiou CF, Stevens SR. Reductions in healthcare resource utilization in psoriatic arthritis patients receiving etanercept therapy: results from the educate trial. J Drugs Dermatol. 2007 Mar;6(3):299-306. PMID 17373192
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com